CLINICAL TRIAL: NCT00150111
Title: B Cell Depletion With the Anti-CD20 Monoclonal Antibody Rituximab in the Treatment of Graves' Disease
Brief Title: Rituximab in the Treatment of Graves' Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 014
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Graves´ Disease; Thyroid Associated Ophthalmopathy
Keywords: Graves disease; thyroid; ophthalmopathy; autoimmunity; B lymphocyte depletion; rituximab; immunization
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy; Thyroid Diseases; Eye Diseases; Autoimmune Diseases | interventions — Methimazole; Rituximab; Immunization

INTERVENTIONS:
Drug: Methimazole
Drug: Rituximab
Biological: Immunization with various vaccines

SUMMARY:
Aim:

In a phase II pilot study encompassing 20 patients with Graves' disease to evaluate the effect of rituximab:

1. Biochemically as assessed by markers of disease activity ( free T4, free T3, TSH, TSH-receptor antibodies, anti-TPO)

DETAILED DESCRIPTION:
Background

Rituximab is a chimeric murine/human anti-CD20 monoclonal antibody which was originally introduced in the clinic years ago for the treatment of malignant lymphomas. The antibody is an IgG1 kappa immunoglobulin containing murine light-and heavy chain variable region sequences and human constant region sequences. The Fab domain of rituximab binds to the CD20 antigen on B lymphocytes. Possible mechanisms of cell lysis include complement-dependent cytotoxicity, antibody-dependent cellular cytotoxicity, and induction of apoptosis.

The mechanism(s) behind the favourable response of rituximab in autoimmune cytopenias are unsettled. A depletion of peripheral blood B cells occurs after just one antibody infusion. Accordingly, it has been proposed that opsonized CD20+ B cells inhibit and saturate macrophage Fc-receptor function and thereby clearance of IgG-coated blood cells by reticuloendothelial cells. Suppression of auto reactive B-cell clones may be another potential mechanism.

Most recently several studies have shown that rituximab- also is very effective in the treatment of various autoimmune cytopenias and autoimmune diseases - idiopathic thrombocytopenic purpura (ITP), warm and cold autoimmune haemolytic anemias, autoimmune neutropenia, pure red cell aplasia, Wegener's granulomatosis, systemic lupus erythematosus, membranous glomerulonephritis, and rheumatoid arthritis - , including disorders which have been considered to be primarily diseases elicited by aberrant T-cell responses, e.g., rheumatoid arthritis. However, recently the importance of the B-cell in the pathogenesis of these autoimmune disorders have been debated and emphasized.

Graves' disease is an autoimmune disease in which both B- and T-cells are activated and participate in its pathogenesis. However, B-cell activation with the production of IgG - thyroid-stimulating antibodies, binding to and activating the thyrotropin receptor on thyroid cells is a prerequisite for the development of Graves' hyperthyroidism. The thyroid-stimulating antibodies cause thyroid hypersecretion, hypertrophy and hyperplasia of the thyroid follicles and ultimately diffuse goiter together with clinical hyperthyroidism. In addition to thyroid-stimulating antibodies against thyroglobulin and thyroid peroxidase are also produced in Graves' disease. The pathogenesis of the other clinical features of disease - the ophthalmopathy and the localized dermopathy or myxedema - is far less elucidated. It has been proposed that the ophthalmopathy develops consequent to an autoimmune response to the thyrotropin receptor, which is also expressed by a preadipocyte subpopulation of orbital fibroblasts. The treatment of Graves' disease includes antithyroid drugs, radioactive iodine and surgery. All three treatment modalities are associated with adverse effects or side-effects.

The most serious complication of antithyroid drugs is agranulocytosis and less frequently acute hepatic necrosis, cholestatic hepatitis and vasculitis. As to treatment with radioactive iodine this therapy may worsen ophthalmopathy. In addition, the treatment is followed by hypothyroidism in a large proportion of the patients.

Based upon the above mentioned observations of a very effective response in many patients with otherwise refractory autoimmune disorders and the pathogenetic concept of Graves' disease as a disorder elicited by auto antibodies stimulating the thyrotropin receptor on thyroid cells ( hyperthyroidism and goiter) and similar antigens in the orbit ( ophthalmopathy ) the hypothesis is that B-cell depletion with rituximab may be a very efficacious therapy reducing or abolishing the production of the auto antibodies which are responsible for Graves' disease.

Aim of the study:

In a phase II pilot study encompassing 20 patients with Graves' disease to evaluate the effect of rituximab:

1. Biochemically as assessed by markers of disease activity ( free T4, free T3, TSH, TSH-receptor antibodies, anti-TPO)

Study design

Material and methods 20 patients with recent onset untreated Graves' disease start antithyroid treatment (methimazole). When euthyroidism is reached - defined by normal thyroid parameters (free T4, free T3, and TSH) - the patients are randomised to +/- rituximab treatment.

Afterwards, the 2 patient groups are followed for 1 year:

* 10 euthyroid patients treated 4 weeks with rituximab, when antithyroid treatment is discontinued.
* 10 euthyroid patients who do not receive rituximab antithyroid treatment being discontinued after 4 weeks.

Effect parameters

Differences in relapse, remission rate at 3, 6, 9 and 12 months follow up/ time to relapse as assessed by:

• Biochemistry ( free T4, free T3, TSH, TSH-receptor antibodies, anti-TPO)

Treatment

Rituximab in a dose of 375 mg/m², administered by iv. Infusion once a week for 4 weeks.

Premedication with paracetamol 1g p.o. or tavestin 2 mg i.v. is given 30-60 min. before each infusion.

ELIGIBILITY:
Inclusion Criteria:

* Graves´ disease
* Adequate anticonception in women.

Exclusion Criteria:

* Performance status >2
* Previous rituximab treatment
* Immunosuppressive treatment
* Serious concomitant disease
* Active infections
* Pregnancy / breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-06; Study Completion 2006-10

PRIMARY OUTCOMES:
Time to relapse after cessation of treatment judged at 1, 3, 6, 9 and 12 months post cessation.

SECONDARY OUTCOMES:
Safety
Changes in autoantibodies (monthly)
Immunological changes (monthly)
Response to vaccines (1 month post-immunization)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel El-Fassi, MD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Department of Endocrinology, Odense University Hospital, Odense, Funen
  - Department of Hematology, Odense University Hospital, Odense

REFERENCES:
- [Background] El Fassi D, Nielsen CH, Hasselbalch HC, Hegedus L. The rationale for B lymphocyte depletion in Graves' disease. Monoclonal anti-CD20 antibody therapy as a novel treatment option. Eur J Endocrinol. 2006 May;154(5):623-32. doi: 10.1530/eje.1.02140. PMID 16645007